CLINICAL TRIAL: NCT02315937
Title: Hemodynamic Assessment During Spinal Anesthesia Using Transthoracic Echocardiography'
Acronym: SATE
Status: Suspended | Type: Observational
Why Stopped: logistic reasons; amendment pending with IRB
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Harm Scholten, MD, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL50108.060.14
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hypotension; Hypovolemia
MeSH Terms: conditions — Hypotension; Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: transthoracic echocardiography — measurement of inferior vena cava diameter during inspiration and expiration using transthoracic echocardiography

SUMMARY:
Rationale: Spinal anesthesia is a safe, frequently used anesthetic technique. The main side effect of spinal anesthesia is hypotension, occuring in up to 85 % of selected cases. This hypotension is often treated with fluid infusion. However, especially in elderly patients, high volume fluid infusion can lead to fluid overload.

The effects of spinal anesthesia on preload and fluid responsiveness are not exactly known. Hence, therapy for hypotension after spinal anesthesia might not be adequate. With transthoracic echocardiography, vena cava inferior diameter and collapsibility can be used to monitor fluid responsiveness and guide fluid management.

Objective: This study has two main objectives. The first is to explore the effects of spinal anesthesia on hemodynamic parameters of fluid status, especially vena cava inferior diameter and collapsibility. The second goal is to test the interrater variability transthoracic echocardiography exams when performed by (trained) anesthesiologists.

Furthermore, the correlation between vena cava inferior collapsibility and the occurence and degree of hypotension (defined as a decrease from baseline of >20% or a systolic pressure < 90 mmHg) after spinal anesthesia will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adult age (>18 years)
* Written informed consent
* Minor surgery under the umbilicus, e.g. herniorrhaphy, transurethral resection of bladder or prostate, orthopaedic procedures
* ASA class I or II

Exclusion Criteria:

* No informed consent
* ASA class III or higher
* Obstetric surgery
* Emergency procedures
* Pre-existing neurological injury or disease
* Contra-indications for spinal anesthesia (e.g. coagulation abnormalities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing spinal anesthesia for minor surgery below the umbilicus
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
vena cava inferior collapsibility (in %) | 1 hour
  vena cava inferior collapsibility: (Maximum vena cava inferior diameter - Minimum vena cava diameter)/maximum vena cava diameter

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bouwman, PhD, Study Director — Catharina Ziekenhuis Eindhoven; Harm Scholten, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands